CLINICAL TRIAL: NCT05517252
Title: Effect Of Tele-Yoga On Aerobic Capacity, Respiratory Muscle Strength, And Cognitive Performance In Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Effect Of Tele-Yoga On Aerobic Capacity, Respiratory Muscle Strength, And Cognitive Performance In Patients With OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, FİLİZ EYÜBOĞLU, Lecturer, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UskudarUn
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; yoga; aerobic capacity; respiratory muscle strength; neurocognitive performance
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Tele-Yoga and Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Yoga Group (Experimental): OSAS patients in the Tele-Yoga group will be taken to group-based Hathastyle Tele-Yoga sessions of 60 minutes three times a week for 12 weeks, simultaneously in groups of 4-5 people, in an internet-based telerehabilitation environment.
  Interventions: Other: Tele - Yoga
- Control Group (Experimental): OSAS patients in the control group will be taught unilateral basal and apical chest expansion exercises in the first session and will be followed as a home program. 3-4 thoracic extension exercises and 1-2 breathing control will be repeated 10 times. The patient will be asked to do the home program four times a day and keep a diary for the home program.
  Interventions: Other: Thoracic Expansion Exercise

INTERVENTIONS:
Other: Tele - Yoga — Telehealth interventions with Yoga are called Tele-yoga. Tele-Yoga aims to provide Yoga support to patients at low cost with the same quality and safety as face-to-face
  Arms: Tele-Yoga Group
Other: Thoracic Expansion Exercise — Thoracic expansion exercises are deep breathing exercises that focus on inspiration and help to loosen secretions on the lungs. Inspiration is active and usually combined with a three-second, end-inspiratory hold before a passive, relaxed and unforced expiration.
  Arms: Control Group

SUMMARY:
OSAS has adverse effects on the functional capacity and quality of life of patients. This study aims to examine the impact of yoga on aerobic capacity, respiratory muscle strength, and cognitive performance in patients with OSAS. Patients will be randomly divided into two groups training (yoga) and control groups. The physical and demographic characteristics of the cases who signed the consent form will be recorded. Anthropometric measurements, circumference measurements, respiratory muscle strength (MIP and MEP), six-minute walking test (6MWT), and cardiopulmonary exercise test (CPET) will be performed. Corsi Blocks Touch Test, Continuous Performance Test, and Stroop Test will be applied to evaluate cognitive performance. The Pittsburg Sleep Index will be used for sleep quality, the Epworth Sleepiness Scale for sleepiness, and the SF-36 scales for health-related quality of life. Subjects with OSAS in the yoga group will be included in group-based yoga sessions of 60 minutes, 3 times a week for 12 weeks. Unilateral basal and apical thoracic expansion exercises will be taught to the patients with OSAS in the control group in the first session. They will be followed as a home program. At the end of the sixth and twelfth week, the evaluations will be made again and the result measurements will be taken.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a syndrome characterized by recurrent upper airway obstructions and accompanying a decrease in oxygen saturation during sleep. The prevalence of OSAS is increasing with the aging population and the obesity epidemic. OSAS has adverse effects on the functional capacity and quality of life of patients. This study aims to examine the effect of yoga on aerobic capacity, respiratory muscle strength, and cognitive performance in patients with OSAS. Patients will be randomly divided into two groups training (yoga) and control groups. The physical and demographic characteristics of the cases who signed the consent form will be recorded. Anthropometric measurements, circumference measurements, respiratory muscle strength (MIP and MEP), six-minute walking test (6MWT), and cardiopulmonary exercise test (CPET) will be performed. Corsi Blocks Touch Test, Continuous Performance Test, and Stroop Test will be applied to evaluate cognitive performance. The Pittsburg Sleep Index will be used for sleep quality, the Epworth Sleepiness Scale for sleepiness, and the SF-36 scales for health-related quality of life. Subjects with OSAS in the yoga group will be included in group-based yoga sessions of 60 minutes, 3 times a week for 12 weeks, in groups of 4 to 5 participants, synchronously in live sessions in an internet-based telerehabilitation environment. Yoga sessions will progress according to the protocol determined according to the weeks. Unilateral basal and apical thoracic expansion exercises will be taught to the patients with OSAS in the control group in the first session. They will be followed as a home program. At the end of the sixth and twelfth week, the evaluations will be made again and the result measurements will be taken. Then, the final measurements of the groups will be compared with statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with clinically stable mild, moderate, and severe OSAS.
* Patients who had an internet network connection at home, had or could install a video telephony software program on their phone or computer

Exclusion Criteria:

* Subjects with a history of buccopharyngeal surgery,
* Concomitant severe orthopedic problems,
* Severe heart failure (New York Heart Association Classification III or IV, left ventricular ejection fraction <45%)
* Severe neurologic disease,
* Body mass index > 40 kg/m2,
* Major pulmonary dysfunction or diabetes,
* Uncontrolled hypertension,
* Trauma affecting the upper airways,
* Stroke or myocardial infarction in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Aerobic Capacity | 12 week
  Symptom-limited Cardiopulmonary Exercise Test (CPET) was performed on a treadmill to determine the aerobic capacity of the patients
Cognitive Performance | 12 week
  Corsi Block Tapping Test and Stroop test were performed to measure cognitive function.
Respiratory Muscle Strength | 12 week
  Respiratory muscle strength was measured using an electronic mouth pressure measuring device (Cosmed Ponyy Fx, Rome, Italy). Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) were measured.

SECONDARY OUTCOMES:
Functional Aerobic Capacity | 12 week
  The six-minute walk test (6MWT) was used to assess functional capacity. Patient was asked to walk for six minutes in a 30-meter corridor as fast as possible at his/her own walking pace. Before and after the test, heart rate and SpO2 were measured by pulse oximetry were recorded; blood pressure, and respiratory frequency were measured. At the end of the test, the distance walked by the subject for six minutes was recorded.
Daytime Sleepiness | 12 week
  Epworth Sleepiness Scale (ESS), consisting of eight questions, was used to measure the general sleepiness of the subjects during the day. On the scale, answers for each question are scored between 0 and 3, and a total score is obtained.
Sleep Quality | 12 week
  The Pittsburgh Sleep Quality Index (PSQI) is a scale consisting of 24 questions that provide detailed information about sleep quality and the type and severity of sleep disturbance in the last month
Health-Related Quality Of Life | 12 week
  The Short Form Scale (SF-36) Quality of Life Questionnaire assessed overall health-related quality of life. This questionnaire consists of eight sections: physical functioning, physical role limitations, bodily pain, general health perception, energy/vitality, social functioning, emotional role limitations, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal Ince, Phd, Study Director — Hacettepe University; FİLİZ EYÜBOGLU, MSc, Principal Investigator — Uskudar University; Berna KARAMANCIOGLU, Principal Investigator — Uskudar University; Naciye VARDAR YAGLI, PhD, Principal Investigator — Hacettepe University; Defne KAYA UTLU, PhD, Principal Investigator — Uludag University; Orhan DALKILIC, PhD, Principal Investigator — Hisar Intercontinental Hospital; GOKSEL SOMAY, PhD, Principal Investigator — Intermed Ciftehavuzlar
Locations (1):
- Uskudar University Physiotherapy and Rehabilitation Application and Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No